CLINICAL TRIAL: NCT02218112
Title: Effect of Weight Loss Induced by a Bypass Surgery on Renal Salt Excretion, Renal Hemodynamic and on Neurohormonal Responses During an Induced Orthostatic Stress in Obese Patients
Brief Title: Impact of Weight Loss After a Bypass Surgery on Renal Hemodynamic Under Stress Conditions
Acronym: OBBYSS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, PD Dr. Grégoire Wuerzner, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: SNF_ 32003B_149903
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Bariatric Surgery; Blood Pressure
Keywords: Blood pressure; Obesity; Glomerular filtration rate; Renal Sodium handling
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OB - Bariatric surgery (gastric bypass): Obese patients who will undergo a bariatric surgery (gastric bypass)
  Interventions: Procedure: bariatric surgery (gastric bypass)
- OB- Control group: Obese patients who will not undergo surgery - Control group

INTERVENTIONS:
Procedure: bariatric surgery (gastric bypass)
  Groups: OB - Bariatric surgery (gastric bypass)

SUMMARY:
The sympathetic nervous (SNS) and the renin angiotensin aldosterone system (RAS) have a direct impact on renal hemodynamic, hormonal secretion and vasoactive peptide. Many mechanisms including the SNS, RAS and renal sodium handling could explain the pathogenesis of hypertension in obese patients. Lifestyle changes and bariatric surgery induce weight loss, which is associated with blood pressure lowering in obese patients. A diminution in the renal sympathetic stimulation and RAS activation could explain this effect.

The AIM of this study is to show that weight loss induced by bypass surgery in obese patients affects renal salt excretion under " low body negative pressure (LBNP)" conditions .

Secondary objectives are to investigate the impact of weight loss on renal hemodynamic (glomerular filtration rate (GFR), renal plasma flow) and neurohormonal responses under " low body negative pressure conditions ". We will also analyse renal blood oxygenation with Blood Oxygenation dependant IRM (BOLD-IRM) technique before and after weight loss.

The population of this study will consist in two groups including 36 patients. The first one will include 24 obese patients that are going to undergo a bariatric surgery. The second one will include 12 obese patients without any weight loss associated surgery.

Both group will undergo 3 investigation days. Each patient will have to undergo a screening visit that will provide dietary advice to ensure a standardized salt intake (120-180 mmol/day) for the duration of the study. The first investigation will define baseline, the second and third day of investigation will take place after 3 month and 12 month after bariatric surgery for surgical patients or after baseline for patients without surgery. One to two weeks before phase 1 and 3 patients will perform a BOLD-MRI. The surgery group will undergo bariatric surgery between the first investigation phase (baseline) and the second. An ambulatory blood pressure and 24-hour urine collection will precede each investigation day. An investigation day consists in renal hemodynamics, neurohormonal and natriuretic response measurements before, during and after 60 min of LBNP at -30mbar . The duration of the study per subject is going to take 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI >35 Kg/m2
* Understanding and signing the informed consent
* Estimated glomerular filtration rate >60 ml/min/1.73 m2

Exclusion Criteria:

* Acute disease
* Asthma or history of asthma
* Patient participating in another clinical trial 30 days before the beginning of the study
* Blood donation (450ml) 2 months before the beginning of the study
* Chronic medication which influence renal function (NSAIDS, Others)
* Allergy
* Documented renal arterial stenosis
* History of symptomatic orthostatic hypotension
* Kidney transplantation
* Kidney malformation / polycystic kidney disease
* Impaired judgement
* Liver failure with ascitis
* Hip circumference at the upper anterior iliac spine > 130cm
* Waist circumference >180cm and weighing > 220kg
* Contraindication/Allergy to furosemide, PAH or Inulin
* Contraindication to MRI if the patient is going to undergo BOLD-MRI
* Postprandial glycemia > 11.0 mmol/L in diabetic patients
* Blood pressure > 180/110 assessed by 24 hour blood pressure measurement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient will briefly be informed about the study during their follow-up at the obesity consultation (Medical Universitary Polyclinic) and the they will be recruited at the Nephrology center in CHUV (Lausanne).
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in sodium excretion | up to one year
  Change in sodium excretion during LBNP conditions

SECONDARY OUTCOMES:
Blood pressure, renal hemodynamic and neurohormonal response | up to one year
  * 24 hour blood pressure measurement
  * Inulin clearance for GFR measurement
  * Renal plasma flow measured with p-aminohippuric acid (PAH) administration
  * Renin plasmatic activity
  * Aldosterone (plasma)
  * Leptin (plasma)
  * Adiponectin (plasma)
  * Plasmatic and urinary electrolytes
  * Plasmatic and urinary lithium

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Zahnd J, Vakilzadeh N, Schwotzer N, Hendriks-Balk M, Mantziari S, Sauser J, Maillard M, Grouzmann E, Favre L, Wuerzner G. Weight loss following gastric bypass increases aldosterone reactivity to orthostatic stress in patients with obesity. Blood Press. 2025 Dec;34(1):2555452. doi: 10.1080/08037051.2025.2555452. Epub 2025 Sep 16. PMID 40892437
- [Derived] Berney M, Vakilzadeh N, Maillard M, Faouzi M, Grouzmann E, Bonny O, Favre L, Wuerzner G. Bariatric Surgery Induces a Differential Effect on Plasma Aldosterone in Comparison to Dietary Advice Alone. Front Endocrinol (Lausanne). 2021 Oct 5;12:745045. doi: 10.3389/fendo.2021.745045. eCollection 2021. PMID 34675881